CLINICAL TRIAL: NCT05281068
Title: The Combination of Iguratimod and Danazol Versus Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia: A Randomized, Controlled, Multicenter, Open-label Trial
Brief Title: The Combination of Iguratimod and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); China-Japan Friendship Hospital (Other); Beijing Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP030
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: ITP; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — iguratimod; Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iguratimod and Danazol (Experimental): Iguratimod is given at a dose of 25 mg bid. Danazol is given at 200mg bid for 12 weeks.
  Interventions: Drug: Iguratimod; Drug: Danazol
- Danazol (Active Comparator): Danazol is given at 200mg bid for 12 weeks.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Iguratimod — Oral iguratimod (25 mg twice daily) for 12 weeks. Iguratimod is a new drug for the treatment of rheumatoid arthritis (RA) and osteoarthritis (OA), which was filed for marketing in Japan in 2003. It can significantly reduce the inflammatory response, not only selectively inhibit COX-2, but also inhibit the production of inflammatory cytokines, tumor necrosis factor, lymphocytes and immunoglobulins, and has an autoimmunomodulatory effect; it has a rapid onset of action, better efficacy and fewer adverse effects than existing drugs, and is effective in patients for whom other drugs are ineffective. It has been reported in the literature that in vitro iguratimod can inhibit the activity of nuclear factor-κB (NF-κB), which in turn inhibits the production of inflammatory cytokines (interleukin-1, interleukin-6, interleukin-8, tumor necrosis factor alpha). Iguratimod also interacts directly with mouse and human B cells in vitro to inhibit the production of immunoglobulins.
  Other Names: Iremod
  Arms: Iguratimod and Danazol
Drug: Danazol — Oral danazol (200 mg twice daily) for 12 weeks.

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of combination of iguratimod and danazol versus danazol for the treatment of adults with steroid-resistant/ relapse immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 100 adults with steroid-resistant/ relapse ITP in China. Patients were randomized to Iguratimod plus danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×109/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* 18 years older;

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* Congestive heart failure
* Severe arrhythmia
* Nursing or pregnant women
* Aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
* Creatinine or serum bilirubin levels each 1•5 times or more than the normal range
* Active or previous malignancy
* Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up. Interim analysis was scheduled at 50% through recruitment.

SECONDARY OUTCOMES:
Complete remission | 6 months
  The number of participants (responders) with platelet count>=100x10^9/L (CR) and the absence of bleeding.
Partial remission | 6 months
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) without the administration of any other platelet increasing therapy.
Time to response | 6 months
  Time to response was defined as the time from starting treatment to the time to achieve the response.
Duration of response | 6 months
  Duration of response was measured from the achievement of response to the loss of response.
Incidence of treatment-emergent adverse events | 6 months
  Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Institute of Hematology, National Clinical Research Center for Hematologic Disease, Beijing Key Laboratory of Hematopoietic Stem Cell Transplantation, Collaborative Innovation Center of Hematology
Locations (2):
- China (2):
  - Zhuo-Yu An, Beijing
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing